CLINICAL TRIAL: NCT05256498
Title: Electrophysiological Studies of the Human Pudendal Nerve Using Short-duration Extracorporeal Stimulation
Brief Title: AURA 1: Augmenting Urinary Reflex Activity: Study 1
Acronym: AURA1
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Merged with other study
Sponsor: Amber Therapeutics Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Amber AURA1
Record Dates: First submitted 2022-01-24; First posted 2022-02-25 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Overactive Bladder; Urge Incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Amber UI Stimulation (Experimental): Short-duration pudendal nerve stimulation
  Interventions: Device: Picostim Amber

INTERVENTIONS:
Device: Picostim Amber — Picostim Amber temporary (24h) lead placement and extracorporeal stimulation

SUMMARY:
AURA 1 (Augmenting Urinary Reflex Activity: study 1) is a study that evaluates the electrophysiological responses of pudendal nerve stimulation using short-duration extracorporeal stimulation

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged ≥ 18 years with urological indications (OAB, UUI, UFS, retention syndromes and pain)
* Meeting criteria for routine SNM (primary or revision surgery) at the discretion of their normal care urologist.
* Ability and willingness to give informed consent
* Willingness to stay overnight in hospital after SNM procedure (as per routine care)

Exclusion Criteria:

* Patient is pregnant, breastfeeding, or plans to become pregnant during the course of the study (pregnancy tests provided in schedule) [this is an exclusion for SNM in any case]
* Any significant medical condition that is likely to interfere with study procedures, device operation, or likely to confound evaluation of study endpoints
* Any psychiatric or personality disorder at the discretion of the study physician
* Any neurological condition that may interfere with normal bladder function (e.g., stroke, multiple sclerosis, Parkinson's disease; clinically significant peripheral neuropathy, or complete spinal cord injury)
* Patient has uncontrolled type I or type II diabetes as defined by their routine care clinician or diabetes with peripheral nerve involvement
* Patient has history of other non-pelvic neoplasia within 5 years prior to enrolment, except for a cancer that was determined to be local occurrence only, such as basal cell carcinoma, or is receiving or planning to receive anti-cancer or anti-angiogenic drugs
* Patient has proven major autoimmune disease, e.g. scleroderma or immunodeficiency (including use of biologic immunomodulatory drugs at time of procedure)
* Patient is not suitable for the study as determined by their routine care physician for any other reason
* Patient is enrolled in another interventional study excepting observational studies, e.g. SNM registries or in relation to disease (see below)
* Patient participation in vigorous sporting activities where these cannot be restricted for a period of 24h while the extracorporeal lead is in situ.

Specific urological

• As per routine clinical SNM criteria (see: https://www.nice.org.uk/guidance/ipg6434)

Specific technical

* Patient is significantly obese (defined as BMI ≥ 35) so as to limit electrode lead placement using standard approaches
* Skin, orthopaedic or neurological anatomical limitations that could prevent successful placement of the electrode lead
* Subject with a documented history of allergic response to titanium, zirconia, polyurethane, epoxy, or silicone

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Intraoperative pelvic floor electromyography (EMG) | 24 Hours
  Intra-operative measurements of amplitude of pelvic floor EMG upon pudendal nerve stimulation

SECONDARY OUTCOMES:
Pelvic floor electromyography (EMG) | 24 Hours
  Amplitude pelvic floor EMG upon pudendal nerve stimulation
Technical outcomes | 24 Hours
  Number of successfully implanted leads

IPD SHARING:
Plan to Share IPD: No